CLINICAL TRIAL: NCT05227235
Title: 3D Telemedicine: Randomised Controlled Trial
Brief Title: Clinical Trial of 3D Telemedicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Strathclyde (Other); Microsoft Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: INGN22SG035
Record Dates: First submitted 2022-02-02; First posted 2022-02-07 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Telemedicine; Surgery

STUDY DESIGN:
Intervention Model Description: The study will use a combination of within-subjects design (crossover) and between-subjects design (standard randomised controlled trial with 2 arms).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of Telemedicine it is not possible to blind the participant (patient) or the care provider (clinician performing consultation). The investigator and outcomes assessor will be blinded, with group allocation blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Telemedicine (Experimental): 3D Telemedicine system allowing patient to be seen in 3 dimensions
  Interventions: Other: 3D Telemedicine
- 2D Telemedicine (Active Comparator): 2D Telemedicine system allowing patient to be seen in standard video call
  Interventions: Other: 2D Telemedicine

INTERVENTIONS:
Other: 3D Telemedicine — Clinical consultation with patient performed with 3D Telemedicine
  Other Names: Telepresence
  Arms: 3D Telemedicine
Other: 2D Telemedicine — Clinical consultation with patient performed with 2D Telemedicine as standard of care
  Other Names: Traditional Telemedicine
  Arms: 2D Telemedicine

SUMMARY:
This randomised controlled trial will provide definitive answers to whether a 3D telemedicine system makes a remote consultation more similar to meeting a doctor face-to-face, than a 2D Telemedicine consultation. This will be measured using a "Presence" scale - which is a measure of the realism or immersion of the system - and is of key importance as preliminary data from the research team's feedback studies found that realism of a clinical consultation correlates strongly with patient satisfaction. Patient satisfaction is seen by many healthcare systems as primary evidence of efficacy of treatment and as a strong determinant of overall health outcomes. Further outcome measures in this trial will assess patient satisfaction, usability, and mental effort.

DETAILED DESCRIPTION:
1. Pre-study Protocol Optimisation Focus group research and co-design with patients from 2019 to 2021, has been used to allow protocol optimisation prior to the RCT. This part of the research project has already been completed by the research team.
2. Pre-study Glasgow Telemedicine Scale Validation Prior to the RCT the research team will validate the Glasgow Telemedicine Scale. This has been developed with experts in digital health, clinicians and patients, and also from the feedback data from previous research. This will involve a group of 20 patients who will attend the Telemedicine clinic and use both the 3D and 2D telemedicine systems without randomisation. Patients who participate in the validation study will complete the questionnaire on their first visit, and return at 6 weeks to use the system again and complete the same questionnaire again.
3. Approach and Design This study will use a randomised crossover design for the primary outcome measure (Single Item Presence Questionnaire). Patients will be randomised to either the 3D or 2D Telemedicine consultation first, and then crossover to the other Telemedicine system. A crossover design has been used in other digital research trials by the research group, as a washout period is not mandatory for tests of perception (such as Presence) as opposed to tests of knowledge. Additionally, plastic surgery patients are known to have a very heterogenous mix of operations and anatomical areas, and a crossover design will account for this heterogeneity better than a between-subjects design. Patients will therefore act as their own controls. Carry-over effects will be analysed in this study. However, to exclude carry-over effects, the study will also analyse the outcome measures between-subjects for the first Telemedicine system used. In these analyses, 2D Telemedicine will be the control group and 3D Telemedicine will be the "intervention" group. The study will be adequately powered to account for within and between subjects outcomes analyses in this trial.

Sample Size Sample sizes were calculated using data from the research team's feedback study of 23 patients performed in 2020-21. For the primary outcome (Single Item Presence Score) at Alpha 0.05 and power 80% a sample size of 9 per group would be required. For the secondary outcome (Telehealth Usability Questionnaire) at Alpha 0.05 and power 80% a sample size of 40 per group would be required. The study will be powered to allow us to assess both primary and secondary outcomes with a between subjects design. Total recruitment will be 80 patients. Given that there is no follow up required by patients and therefore no expected loss to recruitment during the study period, the total recruitment will be the same as the sample size at 80 patients.

Patient Identification Patients will be recruited consecutively from the plastic surgery clinics at the Canniesburn Plastic Surgery Unit, from the sarcoma, plastic surgery and orthoplastic clinics under the care of the PI.

Setting The patient will attend the West Glasgow Ambulatory Care Hospital, Glasgow for the Telemedicine clinic. The clinician will be at a remote location at the Canniesburn Plastic Surgery Outpatient clinic, at Glasgow Royal Infirmary.

Randomisation Process Randomisation will be to 3D or 2D Telemedicine system first. Randomisation will be blocked randomisation of unknown length, generated by computer and held remotely by a password protected system. The research team will collect the randomisation order when the patient attends for the study, once they have completed the consent forms for this study.

Patient Flow in Telemedicine Clinic The patient will be reviewed by the clinician in allocated Telemedicine system 1 for 10 minutes. They will then be reviewed on the same day by the same clinician with Telemedicine system 2 for 10 minutes. The clinician involved will be a Consultant, Training Grade Doctor, Physiotherapist or Nurse Specialist from the Canniesburn Regional Plastic Surgery Unit. A number of clinicians (6 in total) will be used to reduce potential for bias that may arise from using a single consulting clinician. They will be fully trained in the use of the system and the research protocol. The clinical consultation will be standardized between the two systems, to minimize bias. The questions and anatomical areas from the first consultation will be recorded by the clinician using a study Proforma, and used in the second consultation. The patient will subsequently fill in the study questionnaire and complete the exit interview. The patient then requires no further participation in the study.

Data Analysis Statistical analysis will be by independent review by the University of Strathclyde, with results blinded for group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a plastic surgery procedure including:

  * free flap reconstruction
  * pedicled flap reconstruction
  * skin graft reconstruction
  * major cancer surgery
  * major trauma and burns surgery
* Patients able to read and understand English
* Patients able to give informed consent

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* Patients who do not have capacity to consent
* Patients who are registered blind or deaf
* Patients undergoing minor operations only including:

  * primary closure
  * minor local flap reconstruction (for example minor surgery for benign lesions or low risk tumours including Basal or Squamous Cell Carcinoma)
  * minor hand surgery not requiring major flap reconstruction (for example nail bed repair, digital nerve repair, infections).
* Patients with perineal reconstruction given the sensitive area of examination

Ages: 16 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Single Item Presence Questionnaire | 1 day (Single time point post randomization)
  This will ask patients the question "To which extent did you feel present in the virtual clinic, as if you were really there?". This is a single item evaluation of presence validated by Bouchard et al 2004.

SECONDARY OUTCOMES:
Telehealth Usability Questionnaire | 1 day (Single time point post randomization)
  A 21 item validated questionnaire from the University of Pittsburgh on the usability of Telemedicine (Parmanto et al, 2016).
Patient Satisfaction | 1 day (Single time point post randomization)
  Measured on a Visual Analogue Scale between 0-100 (Voutilainen et al. 2016).
Mental Effort Rating Scale | 1 day (Single time point post randomization)
  This is a validated single item scale rated from 0-9, used to assess mental effort during tasks (Paas 1992).
Glasgow Telemedicine Scale. | 1 day (Single time point post randomization)
  As current validated questionnaires are not specifically designed to compare 3D and 2D telemedicine systems, the Glasgow Telemedicine Scale was developed to analyse differences. Currently undergoing validation.

CONTACTS AND LOCATIONS:
Locations (1):
- Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data may be shared on appropriate written request, pending agreement from the entire Research Team.